CLINICAL TRIAL: NCT02543827
Title: Prospective Randomized, Double-blind, Parallel-controlled Versus Placebo in a Polyvalent Sublingual Bacterial Vaccine to 3 Months and 6 Months in Women With RUTI for the Immunomodulatory Efficacy Evaluation, Safety and Clinical Impact
Brief Title: Evaluation of the Efficacy and Safety of MV140
Acronym: MV140
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Inmunotek S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MV140-SLG-003; 2013-001838-17 (EudraCT Number)
Record Dates: First submitted 2015-08-17; First posted 2015-09-07 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Urinary Tract Infection Bacterial
Keywords: Vaccine; Recurrent Urinary Tract Infections (RUTI)
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MV140 I (Experimental): The subjects will receive daily dose of MV140 during 6 months
  Interventions: Biological: MV140
- MV140 II (Experimental): The subjects will receive daily dose of MV140 during 3 months and placebo during 3 months
  Interventions: Biological: MV140; Biological: Placebo
- Placebo (Placebo Comparator): The subjects will receive daily dose of placebo during 6 month
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: MV140 — The subjects will receive daily dose of MV140 during 3 or 6 months
  Arms: MV140 I; MV140 II
Biological: Placebo — The subjects will receive daily dose of placebo during 3 or 6 months
  Arms: MV140 II; Placebo

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of a biological vaccine (MV140) in women with Recurrent Urinary Tract Infections (RUTI) compared with a placebo group.

DETAILED DESCRIPTION:
Double blind parallel placebo controlled study. The subjects will receive medication during three or six months and will be followed up during another twelve months.

ELIGIBILITY:
Inclusion Criteria:

* Women who gave their informed consent.
* Age between 18 and 75 years.
* Must be able to meet the dosage regimen.
* Subjects who had had at least 5 episodes of cystitis in the last 12 months.
* Subjects who had not responded to hygienic-sanitary measures and / or suppressive treatment and / or postcoital prophylaxis.
* Subjects who were free of urinary tract infections at the time of inclusion in the study.

Exclusion Criteria:

* Had not given their informed consent.
* Age was not within the established age range.
* Could not offer cooperation and/or had severe psychiatric disorders.
* Presented a pathologic post-micturition residue.
* Presented moderate to severe incontinence.
* Presented genital tumours.
* Presented Urinary tract tumours.
* Presented lithiasis.
* Presented alterations in the immune system.
* Presented complicated UTIs.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Decrease in the number of RUTI exacerbations. | 1 year
  Average reduction of RUTI exacerbations

SECONDARY OUTCOMES:
Severity of RUTI exacerbations | 1 year
  Review of RUTI exacerbations episodes severity per patient
First RUTI exacerbation | 1 year
  When takes place the First RUTI exacerbation for every single patient
Medication consumption | 1 year
  Review of medication consumed from the beginning to the end of the RUTI exacerbation
Health resource consumption | 1 year
  Counting the Health resource consumption due to RUTI exacerbation: visits to specialists, telephone calls, analyzes and urocultures
Number of visits to the emergency service | 1 year
  Counting the number of visits to the emergency service due to RUTI exacerbation
Number of hospitalizations due to RUTI exacerbations | 1 year
  Counting the number of hospitalization days due to RUTI exacerbations
Changes from baseline in RUTI Assessment Test | 1 year
  Compare the RUTI Assessment Test results at the beginning and at the end of the trial
Percentage of difference in immunological parameters from baseline to end of the trial | 1 year
  Compare the changes from specific cell proliferation baseline against antigens of the vaccine.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 1 year
  Review of the number of adverse event per patient

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Lorenzo, PhD; MD-prof, Study Director; Isidoro Martín, PhD; MD, Principal Investigator; Alfonso Sánchez, PhD; MD, Principal Investigator; Manuel José Vicente, PhD; MD, Principal Investigator; Stephen Foley, FRCS (Urol), Principal Investigator
Locations (5):
- Spain (4):
  - Centro de Salud Universidad Centro, Salamanca, Castille and León
  - Centro de Salud Capuchinos, Salamanca, Castille and León
  - Hospital Universitario de Salamanca, Salamanca, Castille and León
  - CENTRO DE SALUD de PEÑARANDA, Peñaranda de Bracamonte, Salamanca, Castilla Y LEÓN
- Royal Berkshire Hospital Nhs Foundation Trust, Reading, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lorenzo-Gomez MF, Padilla-Fernandez B, Garcia-Cenador MB, Virseda-Rodriguez AJ, Martin-Garcia I, Sanchez-Escudero A, Vicente-Arroyo MJ, Miron-Canelo JA. Comparison of sublingual therapeutic vaccine with antibiotics for the prophylaxis of recurrent urinary tract infections. Front Cell Infect Microbiol. 2015 Jun 3;5:50. doi: 10.3389/fcimb.2015.00050. eCollection 2015. PMID 26090341
- [Background] Lorenzo Gomez MF, Collazos Robles RE, Virseda Rodriguez AJ, Garcia Cenador MB, Miron Canelo JA, Padilla Fernandez B. Urinary tract infections in women with stress urinary incontinence treated with transobturator suburethral tape and benefit gained from the sublingual polibacterial vaccine. Ther Adv Urol. 2015 Aug;7(4):180-5. doi: 10.1177/1756287215576648. PMID 26445597
- [Background] Lorenzo-Gomez MF, Padilla-Fernandez B, Garcia-Criado FJ, Miron-Canelo JA, Gil-Vicente A, Nieto-Huertos A, Silva-Abuin JM. Evaluation of a therapeutic vaccine for the prevention of recurrent urinary tract infections versus prophylactic treatment with antibiotics. Int Urogynecol J. 2013 Jan;24(1):127-34. doi: 10.1007/s00192-012-1853-5. Epub 2012 Jul 18. PMID 22806485
- [Background] Sanchez Ramon S, Manzanares M, Candelas G. MUCOSAL anti-infections vaccines: Beyond conventional vaccines. Reumatol Clin (Engl Ed). 2020 Jan-Feb;16(1):49-55. doi: 10.1016/j.reuma.2018.10.012. Epub 2018 Dec 7. English, Spanish. PMID 30527360
- [Background] Sanchez-Ramon S, Perez de Diego R, Dieli-Crimi R, Subiza JL. Extending the clinical horizons of mucosal bacterial vaccines: current evidence and future prospects. Curr Drug Targets. 2014;15(12):1132-43. doi: 10.2174/1389450115666141020160705. PMID 25330031
- [Background] Benito-Villalvilla C, Cirauqui C, Diez-Rivero CM, Casanovas M, Subiza JL, Palomares O. MV140, a sublingual polyvalent bacterial preparation to treat recurrent urinary tract infections, licenses human dendritic cells for generating Th1, Th17, and IL-10 responses via Syk and MyD88. Mucosal Immunol. 2017 Jul;10(4):924-935. doi: 10.1038/mi.2016.112. Epub 2016 Dec 14. PMID 27966556
- [Background] Martin-Cruz L, Sevilla-Ortega C, Benito-Villalvilla C, Diez-Rivero CM, Sanchez-Ramon S, Subiza JL, Palomares O. A Combination of Polybacterial MV140 and Candida albicans V132 as a Potential Novel Trained Immunity-Based Vaccine for Genitourinary Tract Infections. Front Immunol. 2021 Jan 21;11:612269. doi: 10.3389/fimmu.2020.612269. eCollection 2020. PMID 33552074
- [Background] Yang B, Foley S. First experience in the UK of treating women with recurrent urinary tract infections with the bacterial vaccine Uromune(R). BJU Int. 2018 Feb;121(2):289-292. doi: 10.1111/bju.14067. Epub 2017 Nov 23. PMID 29171130
- [Derived] Lorenzo-Gomez MF, Foley S, Nickel JC, Garcia-Cenador MB, Padilla-Fernandez BY, Gonzalez-Casado I, Martinez-Huelamo M, Yang B, Blick C, Ferreira F, Caballero R, Saz-Leal P, Casanovas M. Sublingual MV140 for Prevention of Recurrent Urinary Tract Infections. NEJM Evid. 2022 Apr;1(4):EVIDoa2100018. doi: 10.1056/EVIDoa2100018. Epub 2022 Jan 21. PMID 38319200